CLINICAL TRIAL: NCT05185882
Title: The Effect of Different Focusing Methods on Muscle Activity During The Single Leg Squat Movement
Brief Title: The Effect of Different Focusing Methods on Muscle Activity
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assistant Professor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 2021-388
Record Dates: First submitted 2021-12-04; First posted 2022-01-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Knee Injuries and Disorders
Keywords: single leg squat; muscular activity; knee alignment
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: 1. Single leg squat without a clue or focusing method
  2. Single leg squat with an external focus
  3. Sinlge leg squat with an internal focus
  Interventions: Other: Single leg squat

INTERVENTIONS:
Other: Single leg squat — Single leg squat exercise in different circumstances

SUMMARY:
The aim of this study is to compare the effects of different focusing methods on muscular activity

DETAILED DESCRIPTION:
After the first data collecting ( Demographic data, Inclusion criteria) surface electromyography EMG evaluations will be taken from 6 muscles( Vastus Medialis, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Semitendinosus, Gluteus Medius). These recordings will be taken in 3 different circumstances: 1- Without a focusing method 2- With an external focus and 3- With an internal focus

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Having a Body Mass Index between 18.5-24.9

Exclusion Criteria:

* Having trauma/surgery involving the lower extremity in the last 6 months or having any disorder affecting hip and knee muscle function
* Foot Posture Index score not being between 0 and +5
* Hamstring Flexibility- Sit and Reach Test score greater than +5 cm
* Restricted ankle dorsiflexion angle (It will be expected to be at least 5 degrees more than neutral)

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography | Procedure (During the intervention)
  Surface EMG evaluations of Vastus Medialis, Vastus Lateralis, Rectus Femoris, Biceps Femoris, Semitendinosus and Gluteus Medius Muscles in 3 conditions in a row(Without a focusing method, With an internal focus, With an external focus

SECONDARY OUTCOMES:
Foot Posture Index | Baseline, for inclusion criteria
  Evaluations of Foot by inspection
Sit and Reach Test | Baseline, for inclusion criteria
  Assessment of hamstring flexibility
Gluteus Medius Muscle Dynamometer Assessment | Baseline, for inclusion criteria
  Assessment of Gluteus Medius Strength
Ankle Dorsi Flexion Goniometer Assessment | Baseline, for inclusion criteria
  Assessment of Dorsiflexion

CONTACTS AND LOCATIONS:
Overall Officials: Emre Serdar Atalay, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Emre Serdar Atalay, Ankara, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No